CLINICAL TRIAL: NCT06706011
Title: Swedish Title: Virtuella Patienter - en Interaktiv Utbildningsmodul Inom Universitet Och högskola. In English: Virtual Patients - An Interactive Educational Module in Universities and Colleges.
Brief Title: Virtual Patients - An Interactive Educational Module for Higher Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Karolina Sörman, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023-06687-01
Record Dates: First submitted 2024-10-28; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Psychiatric Problem; Psychiatric Issue; Violence
Keywords: virtual patient; education

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Virtuel Patient
  Interventions: Other: Virtual Patient
- Control (No Intervention): No Virtuel Patient

INTERVENTIONS:
Other: Virtual Patient — Interactive Educational Activity
  Arms: Intervention

SUMMARY:
Popular Science Summary (for the whole project)

In modern healthcare, several challenges exist: short patient visits, highly specialized care, and limited opportunities for education and professional development among healthcare staff. In theoretical training efforts, it can be difficult to highlight and provide opportunities to practice complex patient interactions. The overall goal of this project is to evaluate the effects of an interactive educational module that includes training with virtual patients (VP). Single training sessions rarely lead to behavioral changes in clinical practice, but concrete training with a clear connection to clinical tasks can have a better effect.

In this research project, VPs will be part of an educational module at universities and colleges, where the overarching goal is for students to practice clinically relevant communication areas. Two main areas have been selected for the VP in this project: intimate partner violence and suicide risk assessment. Both of these areas are of great significance to public health and have direct relevance to clinical care, especially in psychiatry. Specific objectives of the project include exploring the user experience of the VP, examining whether the VP contributes to increased knowledge and confidence in asking questions within the chosen focus area, studying students' experiences of using the VP, how it has influenced their work with patients after graduation, and finally, examining user patterns on the VP platform.

Previous research suggests that virtual patient cases can have positive effects on learning and engagement and may even be more effective than traditional education in improving clinical decision-making and critical thinking skills. VPs have been studied in various medical specialties, but there is a lack of knowledge specifically in psychiatry. In this project, researchers will evaluate the use of VPs in psychiatric training within medical, nursing, and psychology programs.

DETAILED DESCRIPTION:
Overall purpose (for the whole project):

To investigate virtual patient cases (VP) as an interactive educational module for students in universities and colleges. The educational module will consist of three parts: a theoretical and preparatory lecture, training with VP, and a follow-up seminar. The aim is to evaluate how well this module prepares students to ask clinically relevant questions in focus areas such as intimate partner violence and suicide risk assessment. The target group for the project is students in nursing, medical, and psychology programs at various universities and colleges in Sweden.

Specific aims for this study:

To investigate whether VP contributes to an increased level of knowledge and confidence in asking questions within the selected focus areas among students in nursing, medical, and psychology programs.

Focus areas for VP:

Intimate partner violence

ELIGIBILITY:
Inclusion Criteria:

* Students in Nursing Program

Exclusion Criteria:

* None, except if the student does not want to participate

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2024-08-26 (Actual); Primary Completion 2024-09-09 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
General Self-Efficacy Scale | Up to two months
  This scale is a self-report measure of self-efficacy. Likert scale 1-4: 1=Not at all true, 2=Hardly true, 3=Moderately true, 4=Exactly true.
General Self-Efficacy - Visual Analog Scale | Up to two months
  Measuring self-efficacy. Scale 1-10: 1=Low, 10=High.
Level of Knowledge - Test | Up to two months
  Measuring level of knowledge. 15 multiple-choice question about inpartner violence.
Level of Knowledge - Visual Analog Scale | Up to two months
  Measuring level of knowledge, Scale 1-10: 1=Low, 10=High.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Psychatry Research, Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No